CLINICAL TRIAL: NCT02182310
Title: Assessment of the Effect of 480 mg and 1200 mg of BI 201335 as Single Dose on the QT Interval in Healthy Female and Male Subjects. A Randomised, Placebo Controlled, Double-blind, Four-way Crossover Phase-I-study With Moxifloxacin as Positive Control
Brief Title: Assessment of the Effect of BI 201335 on the QT Interval in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.16
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — faldaprevir; Moxifloxacin

ARMS (5):
- BI 201335 placebo (Placebo Comparator): crossover part
  Interventions: Drug: BI 201335 placebo
- BI 201335 low dose (Experimental): crossover part
  Interventions: Drug: BI 201335 low dose
- BI 201335 high dose (Experimental): crossover part
  Interventions: Drug: BI 201335 high dose
- Moxifloxacin (Active Comparator): crossover part
  Interventions: Drug: Moxifloxacin
- BI 201335 or Placebo (Experimental): tolerability part in female subjects
  Interventions: Drug: BI 201335 placebo; Drug: BI 201335 high dose

INTERVENTIONS:
Drug: BI 201335 low dose
  Arms: BI 201335 low dose
Drug: BI 201335 placebo
  Arms: BI 201335 or Placebo; BI 201335 placebo
Drug: Moxifloxacin
  Arms: Moxifloxacin
Drug: BI 201335 high dose
  Arms: BI 201335 high dose; BI 201335 or Placebo

SUMMARY:
To demonstrate that BI 201335 does not prolong the QT interval more than placebo.

To assess the tolerability of 1200 mg of BI 201335 as single dose in female subjects (double-blind, randomised, placebo-controlled) before inclusion of female subjects in the cross-over part of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian males and females, 18 to 50 years of age
* Body mass index (BMI) ranging from 18.5 to 29.9 kg/m2 (BMI calculation: weight in kilograms divided by the square of height in meters)
* Signed written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ 30 days prior to administration or during the trial)
* Heavy smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any deviation of a laboratory value that is considered to be of clinical relevance
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to BI 201335, moxifloxacin or related drugs of these classes
* Homozygous genotype status for "Gilbert" polymorphisms (Uridine diphosphate (UDP)-glucuronosyl transferase 1A1 (UGT1A1)*28, *60)
* Heart rate at screening of > 85 bpm or < 40 bpm
* Any screening ECG value outside of the reference range of clinical relevance including, but not limited to pulse rate (PR) interval > 220 ms, QRS interval > 115 ms, QTcB (QT interval, corrected for heart rate according to Bazett's formula) > 470 ms, or QT (uncorrected) > 470 ms
* For Female subjects

  * Pregnancy
  * Positive pregnancy test
  * No adequate contraception (adequate contraception e.g. sterilisation, intrauterine pressure , oral contraceptives). Females, who are not surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)
  * Inability to maintain this adequate contraception during the whole study period from the time of screening until one month after the last intake
  * Lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
QTcI interval (QT interval individually corrected for heart rate) | pre-dose and 3 to 8 hours

SECONDARY OUTCOMES:
The mean value of QTcI changes from baseline between 2 h and 24 h after dosing | Pre dose and 2 to 24 hours post dosing
The change from mean baseline of the QTcI at any point in time between 2 h and 24 h after dosing | Pre dose and 2 to 24 hours post dosing
The time-matched changes versus placebo in QTcI at any point in time between 2 h and 24 h after dosing | Pre dose and 2 to 24 hours post dosing